CLINICAL TRIAL: NCT02301819
Title: ExtraCorporeal Membrane Oxygenation in the Therapy of Cardiogenic Shock
Acronym: ECMO-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Na Homolce Hospital (Other)
Collaborators: General University Hospital, Prague (Other); University Hospital Pilsen (Other)
Responsible Party: Principal Investigator, Petr Ostadal, Dr., Na Homolce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-5-14 V2
Record Dates: First submitted 2014-11-23; First posted 2014-11-26 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Invasive (Active Comparator): Immediate veno-arterial extracorporeal membrane oxygenation (ECMO)
  Interventions: Device: Veno-arterial extracorporeal membrane oxygenation (ECMO)
- Conservative (Active Comparator): Early conservative therapy according to standard practice
  Interventions: Other: Early conservative therapy according to standard practice

INTERVENTIONS:
Device: Veno-arterial extracorporeal membrane oxygenation (ECMO) — Veno-arterial extracorporeal membrane oxygenation (ECMO) will be ineserted as soon as possible and set to achieve adequate organ and tissue perfusion.
  Arms: Invasive
Other: Early conservative therapy according to standard practice — Standard therapy including inotropes and vasopressors will be used to achieve hemodynamic stabilization and adequate tissue perfusion.
  Arms: Conservative

SUMMARY:
Eligible patients with severe cardiogenic shock will be randomized to one of the two arms: immediate ECMO therapy or early conservative therapy. In the invasive group, veno-arterial ECMO will be implanted according to the local practice with flow settings to ensure sufficient tissue perfusion. With the exception of ECMO implantation in the invasive group, all other diagnostic and therapeutic procedures will be done according to the current standard of care at the tertiary cardiovascular center, including other cardiovascular interventions (i.e. percutaneous coronary intervention or cardiac surgery). Implantation of other mechanical support devices including ECMO in the primary conservative group is allowed in the case of shock progression with rise of serum lactate by 3 mmol/L in comparison with the lowest value during the past 24 hours. Follow-up include visits at 30 days, 6 moths and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfil criteria for rapidly deteriorating (A) or severe (B) cardiogenic shock:

A. Rapidly deteriorating cardiogenic shock is defined as progressive hemodynamic instability necessitating repeated bolus administration of vasopressors to maintain mean arterial pressure > 50 mmHg + impaired left ventricle systolic function (Left ventricle ejection fraction (LVEF) < 35% or LVEF 35-55% in case of severe mitral regurgitation or aortic stenosis) or

B. In severe cardiogenic shock all following criteria should be met:

1. Hemodynamic:

   Cardiac Index (CI) < 2.2 L/min/m2 + norepinephrine dose > 0.1 μg/kg/min + dobutamin dose > 5 μg/kg/min or Systolic blood pressure < 100 mmHg + norepinephrine dose > 0.2 μg/kg/min + dobutamin dose > 5 μg/kg/min + (LVEF < 35% or LVEF 35-55% + severe mitral regurgitation or aortic stenosis)
2. Metabolic:

   Lactate - two consecutive values ≥ 3 mmol/L (with at least 30 min between samples), with non-decreasing trend on steady doses of inotropes and/or vasopressors or SvO2 - two consecutive values < 50% (with at least 30 min between measurements), with non-increasing trend on steady doses of inotropes and/or vasopressors
3. Hypovolemia must be excluded:

Central venous pressure > 7 mmHg or pulmonary capillary wedge pressure > 12 mmHg

Exclusion Criteria:

1. Age < 18 years
2. Life expectancy lower than 1 year
3. High suspicion of pulmonary emboli or cardiac tamponade as a cause of shock
4. Significant bradycardia or tachycardia which might be responsible for hemodynamic instability and not treated by pacing or cardioversion
5. Cardiac arrest survivors remaining comatose
6. Hypertrophic obstructive cardiomyopathy
7. Peripheral artery disease disabling insertion of outflow cannula to femoral artery
8. Moderate to severe aortic regurgitation
9. Aortic dissection
10. Uncontrolled bleeding or TIMI major bleeding within last 6 months
11. Known encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-09; Primary Completion 2022-08 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Composite of death from any cause, resuscitated circulatory arrest, and implantation of another mechanical circulatory support device | 30 days

SECONDARY OUTCOMES:
All-cause mortality | 30 days
All-cause mortality | 6 months
All-cause mortality | 12 months
Neurological outcome (according to Cerebral Performance Category scale) | 30 days

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - Na Homolce Hospital, Prague, Select One
  - Regional Hospital Liberec, Liberec
  - University Hospital Pilsen, Pilsen
  - General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ostadal P, Rokyta R, Kruger A, Vondrakova D, Janotka M, Smid O, Smalcova J, Hromadka M, Linhart A, Belohlavek J. Extra corporeal membrane oxygenation in the therapy of cardiogenic shock (ECMO-CS): rationale and design of the multicenter randomized trial. Eur J Heart Fail. 2017 May;19 Suppl 2:124-127. doi: 10.1002/ejhf.857. PMID 28470919
- [Result] Ostadal P, Rokyta R, Karasek J, Kruger A, Vondrakova D, Janotka M, Naar J, Smalcova J, Hubatova M, Hromadka M, Volovar S, Seyfrydova M, Jarkovsky J, Svoboda M, Linhart A, Belohlavek J; ECMO-CS Investigators. Extracorporeal Membrane Oxygenation in the Therapy of Cardiogenic Shock: Results of the ECMO-CS Randomized Clinical Trial. Circulation. 2023 Feb 7;147(6):454-464. doi: 10.1161/CIRCULATIONAHA.122.062949. Epub 2022 Nov 6. PMID 36335478
- [Derived] Ostadal P, Vondrakova D, Rokyta R, Karasek J, Kruger A, Janotka M, Naar J, Smalcova J, Hubatova M, Hromadka M, Volovar S, Seyfrydova M, Linhart A, Belohlavek J. Cardiac index, SvO2 or pCO2 gap may determine benefit from ECMO in cardiogenic shock: post-hoc analysis of the multicenter, randomized ECMO-CS trial. Crit Care. 2025 Jul 14;29(1):303. doi: 10.1186/s13054-025-05513-5. PMID 40660350